CLINICAL TRIAL: NCT02081573
Title: Brief CBT Interventions Delivered by Nurse Care Managers to Improve Type 2 Diabetes Outcomes: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Judith A. Callan PhD. RN, Research Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13050427; School of Nursing eHub pilot (Other: University of Pittsburgh School of Nursing)
Record Dates: First submitted 2014-03-03; First posted 2014-03-07 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Brief CBT; smartphone app; mHealth; diabetes distress; adherence; cognitive behavioral therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief CBT (Experimental): During the course of the twice/month diabetes management phone sessions the nurse care manager will work collaboratively with the patient to identify a dysfunctional belief that may be affecting adherence and could be improved by a brief CBT intervention (5-7 minutes). The care manager will utilize the CBT phone app to identify a CBT intervention that will be most appropriate for the situation. Each intervention is described step by step in the app. The nurse will go through the intervention and when completed will assure the patient's understanding.CBT interventions are geared towards helping the patient identify and restructure thinking that is impairing successful self-management of a chronic disease
  Interventions: Behavioral: Brief CBT

INTERVENTIONS:
Behavioral: Brief CBT — During the course of the twice/month diabetes management phone sessions the nurse care manager will work collaboratively with the patient to identify a dysfunctional belief that may be affecting adherence and could be improved by a brief CBT intervention (5-7 minutes). The care manager will utilize the CBT phone app to identify a CBT intervention that will be most appropriate for the situation. Each intervention is described step by step in the app. The nurse will go through the intervention and when completed will assure the patient's understanding.CBT interventions are geared towards helping the patient identify and restructure thinking that is impairing successful self-management of a chronic disease
  Other Names: CBT MobileWork

SUMMARY:
Primary aim: examine feasibility and acceptability of a brief cognitive therapy protocol for type II diabetes administered by nurse care managers or health coaches via phone.

DETAILED DESCRIPTION:
A significant problem in primary care healthcare delivery is the lack of interventions to improve medication and overall regimen adherence in persons with Type 2 diabetes (T2DM). Diabetes distress, a negative response to the diagnosis of T2DM, danger of complications, and self-management burdens is present in up to 70% of persons with T2DM. Distress is a significant factor in medication nonadherence and poor glycemic control. Treatment adherence is vital to maintain glucose control and reduce complications.

The literature has identified dysfunctional thinking patterns such as beliefs (e.g., I can't handle taking these medications), assumptions (e.g., I know I will have side effects to these medications) and interpretations (e.g., I'm too overwhelmed to do all of this stuff) as critical variables that impact both distress and T2DM treatment adherence. Current treatment strategies within primary care do not address the dysfunctional thinking patterns that affect the patient's distress level, T2DM medication adherence, and complex daily self-care activities.

Cognitive behavior therapy (CBT), a well-established evidenced-based treatment, helps patients to identify, and restructure dysfunctional thinking patterns. We propose to test a brief CBT approach delivered by nurse care managers and supported by a comprehensive mobile phone CBT skills practice application (app) within primary care. The promising results of our preliminary studies using a mobile phone app to stimulate real-time CBT skills practice prompt us to propose a pilot of its use with patients with T2DM with the following aims:

Primary aim: examine feasibility and acceptability of the assessment protocol, and the recruitment, and retention of study participants.

Secondary aim: 1) collect preliminary data on the effect of the intervention on clinical outcomes, e.g., self-reported adherence to medication and self-management adherence, e.g., diet, exercise; levels of diabetes distress, diabetes medication beliefs, and distal T2DM outcomes (HbA1c level and body mass index).

ELIGIBILITY:
Inclusion Criteria:

Ten adults will be recruited through the UPMC health plan and are treated at a primary care center. To be considered for inclusion subjects must:

1. have a diagnosis of T2DM;
2. have a score of >3 on the Diabetes Distress Scale;
3. be taking at least one oral antihyperglycemic agent (the patient may also be using injectable antihyperglycemic medications, including insulin);
4. have an HbA1c level of greater than 8 at baseline;
5. be receiving treatment for T2DM in the primary care setting;
6. be aged 30 - 65 years and
7. be able to read at the 8th-grade level and to provide informed consent.

Four nurse care managers will also be recruited from UPMC Health Care. To be considered they must be employed at UPMC Health Care and

1. Have received the Brief CBT Training that was given in Phase I of this study;
2. Be identified as a RN or a RN who is a diabetes nurse educator; and have Nurse Care Management responsibilities with patients who have Type 2 Diabetes.

Nurses will be excluded from the study if:

1. They did not successfully complete the training in Phase I or
2. Are not Nurse Care Managers at UPMC Health Care. -

Exclusion Criteria:

The following are exclusion criteria:

1. major psychiatric disorder and suicidal risk;
2. dementia or disorders with substantial cognitive impairment. -

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Callan, PhD, RN, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a small sample feasibility study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a existing cases of nurse care managers and health coaches who administered the study intervention. Individuals who were interested and had HbA1C higher than 8.0 were screened.
Pre-assignment Details: Screened to have mean distress over 2.0 and HbA1C of 8 or above via measurements by our tests.
Groups:
- Brief CBT: During the course of the twice/month diabetes management phone sessions, over 3-4 months, the nurse care manager will work collaboratively with the patient to identify a dysfunctional belief that may be affecting adherence and could be improved by a brief CBT intervention (5-7 minutes). The care manager will utilize the CBT phone app to identify a CBT interventions.
Period: Overall Study
Arm/Group | Brief CBT
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 47.7 [36 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
HbA1C [Mean (Standard Deviation); unit: percent] | 9.8 (.9)
Distress (Diabetes Distress Scale) [Mean (Standard Deviation); unit: mean result on scale] — The Brief Diabetes Distress Scale is a 17 item scale assessing distress in managing diabetes. The scale is scored as an average with a potential range from 1 to 6. Scores of 3 or greater are considered indicating stress.
  Fisher, L., Glasgow, R. E., Mullan, J. T., Skaff, M. M., & Polonsky, W. H. (2008). Development of a brief diabetes distress screening instrument. The Annals of Family Medicine, 6(3), 246-252.
  https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2384991/
  mean result on scale | 3.52 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Questionnaire.
Description: The acceptability questionnaire measures feasibility and acceptability of the Brief CBT protocol. Adapted from Lewis JR.: IBM Computer Usability Satisfaction Questionnaires: Psychometric Evaluation and Instructions for Use. International Journal of Human-Computer Interaction 1995; 7 (1):67-78. Scale is scored as a mean and ranges from 1-7. In this adaptation, lower scores are better satisfaction.
Time Frame: 12 weeks
Population: Mean acceptability of the Brief CBT protocol.
Measure: Mean (Standard Deviation); unit: mean of scale items
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
mean of scale items | 2.49 (1.39)

2. Secondary Outcome: Morisky Questionnaire
Description: Brief scale of adherence to medications. Morisky 5 items was used. Mean score presented. Scale range is from 5-13. Lower score is better adherence. Mean change from baseline to 12 weeks is examined.
Time Frame: 12 weeks
Population: Mean change from baseline to 12 weeks.
Measure: Mean (Standard Deviation); unit: mean of scale items
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
mean of scale items | .10 (1.73)

3. Secondary Outcome: Diabetes Distress Scale
Description: Levels of diabetes distress per standardized questionnaire will be measured before intervention and after intervention. Change of mean score is reported. Change in score from baseline to post followup. Lower score means less distress. Scale range is from 1-6. Adapted from Fisher, L., Glasgow, R.E., Mullan, J.T., Skaff, M.M., Polonsky, W.H. (2008) Development of a Brief Diabetes Screening Instrument. Annals of Family Medicine; 6:246-252.
Time Frame: 12 weeks
Population: Change in score from baseline to post followup
Measure: Mean (Standard Deviation); unit: mean of scale items
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
mean of scale items | -.77 (1.35)

4. Secondary Outcome: Medication Beliefs Scale
Description: Change in medication beliefs from before and after intervention. Adapted from Horne, R., Weinman, J., Hankins, M. (1999). The Beliefs About Medicines Questionnaire: The Development and Evaluation of a New Method for Assessing the Cognitive Representation of Medications. Psychology and Health 14: 1-24.
Time Frame: 12 weeks
Arm/Group | Brief CBT
Number analyzed (Participants) | 0

5. Secondary Outcome: HbA1c Level
Description: Change in HbA1c from before to after treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
percentage of glycosylated hemoglobin | -.22 (1.80)

6. Secondary Outcome: Body Mass Index
Description: Change in Body Mass Index from before to after treatment
Time Frame: 12 weeks
Population: Change BMI over time.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Brief CBT
Number analyzed (Participants) | 10
kg/m^2 | -1.22 (1.39)

ADVERSE EVENTS:
Time Frame: during the participant's participation in the study, 12-16 weeks.
Arm/Group | Brief CBT
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This is a pilot feasibility study with small sample (N=10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No